CLINICAL TRIAL: NCT03013946
Title: A Phase III Study Testing the Role of PRoactivE Coaching on PAtient REported Outcome in Advanced or Metastatic Renal Cell Carcinoma Treated With Sunitinib or a Combination of Pembrolizumab + Axitinib or Avelumab + Axitinib in First Line Therapy
Brief Title: Role of PRoactivE Coaching on PAtient REported Outcome in Advanced or Metastatic RCC Treated With Sunitinib or a Combination of Pembrolizumab + Axitinib or Avelumab + Axitinib in First Line Therapy
Acronym: PREPARE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient accrual rate
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Pfizer (Industry); Crolll Gmbh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AIO-NZK-0115/ass; 2016-000399-28 (EudraCT Number)
Record Dates: First submitted 2016-12-14; First posted 2017-01-09 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Renal Cell Carcinoma, Metastatic; Renal Cell Cancer, Recurrent
Keywords: Therapy-Coaching, Quality of Life
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Coaching) (Experimental): Concomitant coaching (24 weeks) Pro-active TEAE (Treatment emergent adverse events) management Cancer therapy according to Standard of Care (SOC) QoL assessments/ primary endpoint FKSI-15
  Interventions: Behavioral: Concomitant coaching
- Arm B (Control) (No Intervention): Re-activeTEAE management (SOC) Cancer therapy according to Standard of Care (SOC) QoL assessments/ primary endpoint FKSI-15

INTERVENTIONS:
Behavioral: Concomitant coaching — The corner stones of the pro-active coaching are as follows:
  * Patient education:
    * Information on nature and severity of treatment emergent AEs
    * information about remedies for TEAEs
    * propagation and explanation of tests and treatment decisions
    * Patient instruction on self-care and preventive measures
  * Preemptive AE treatment strategies
  * Supervision of reported ADR severity, ADR mitigation strategies according to recommendations of the PREPARE protocol and cancer treatment modification by treating physician in close collaboration with the coach
  Arms: Arm A (Coaching)

SUMMARY:
The primary objective of the trial is to determine the effect of a 24-week concomitant coaching on patient reported outcomes of patients receiving standard treatment for mRCC with sunitinib or a combination of pembrolizumab + axitinib or avelumab + axitinib in first line therapy.

DETAILED DESCRIPTION:
The goal of our study is to define the benefit of proactive coaching in mRCC, when compared to a reactive approach, which is considered the standard of care.

Patients in the Coaching Arm A will be trained continuously at personal interactions of coach and patient (Face-to Face meetings as well as telephone contacts). The patient is educated on nature and severity of treatment emergent Adverse events (TEAE) of sunitinib or a combination of pembrolizumab + axitinib or avelumab + axitinib in first line therapy.

Quality of Life (QoL) is assessed during sunitinib treatment in both arms (Arm A Coaching and Arm B non Coaching).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization (EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age ≥ 18 years at time of study entry
3. Advanced or metastatic renal cell carcinoma, not amendable to surgery with curative intent, rendering the patient eligible for Tyrosin Kinase Inhibitor (TKI) treatment with sunitinib
4. Intended first-line treatment with sunitinib
5. Documented progressive disease within 6 months prior to study inclusion
6. Patients with measurable disease (at least one uni-dimensionally measurable target lesion by CT-scan or MRI) according to modified Response Evaluation Criteria in Solid Tumors (RECIST 1.1) as well as non-measurable disease are eligible.
7. Prior radiotherapy and surgery are allowed if completed 4 weeks (for minor surgery and palliative radiotherapy for bone pain: 2 weeks) prior to start of treatment and patient recovered from toxic effects.
8. Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
9. Subject is willing to receive additional concomitant coaching and able to comply with the QoL/PRO (patient-reported outcome) assessments specified in the protocol for the duration of the study including scheduled visits, examinations and follow up.

Exclusion Criteria:

1. Any other anti-cancer treatment aside of sunitinib for mRCC (except palliative radiotherapy)
2. Previous malignancy (other than mRCC) which either progresses or requires active treatment.

   Exceptions are: basal cell cancer of the skin, pre-invasive cancer of the cervix, T1a or T1b prostate carcinoma, or superficial bladder tumor [Ta, Tis and T1].
3. CNS metastases, unless local therapy has been completed for at least 3 month and patient does not require the use of steroids.
4. Chronic liver disease with Child-Pugh B or C score
5. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year)
6. Any condition that, in the opinion of the investigator, would interfere with evaluation of the concomitant coaching or QoL assessments or interpretation of patient safety or study results
7. Participation in another clinical study with an investigational product during the last 30 days before inclusion
8. Any previous treatment with a tyrosine kinase inhibitor for metastatic disease. Adjuvant or neoadjuvant therapy for localized disease is permitted, provided that relapse occurred at least 6 months after last exposure
9. Previous enrollment or randomization in the present study (does not include screening failure).
10. Involvement in the planning and/or conduct of the study (applies to both Pfizer staff and/or staff of sponsor and study site)
11. Patient who might be affiliated or otherwise dependent on the sponsor, site or the investigator
12. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities [§ 40 Abs. 1 S. 3 Nr. 4 AMG].
13. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
QoL assessment during sunitinib treatment: questionnaire | 24 weeks from randomization
  Rate of responders to concomitant coaching assessed by the (Functional Assessment of Cancer Therapy-Kidney Symptom Index (FKSI)) FKSI-15 questionnaire.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) according to RECIST 1.1 criteria | up to one year from randomization
  Objective Response Rate (ORR) according to RECIST 1.1 criteria
Overall Survival (OS) | up to 36 months from randomization
  Overall Survival (OS)
progression-free survival (PFS) | up to 36 months from randomization
  progression-free survival (PFS)
Duration of treatment (coaching and cancer treatment) | Coaching: up to 24 weeks from randomization / cancer treatment: up to 36 months from randomization
  Duration of treatment (coaching and cancer treatment)
dose density of sunitinib | 24 weeks from randomization
  dose density of sunitinib
Rate of patients receiving treatment beyond progression | up to 36 months from randomization
  Rate of patients receiving treatment beyond progression
Further cancer treatment | up to 36 months
  Further cancer treatment
Time to first subsequent therapy (TFST) | up to 36 months
  Time to first subsequent therapy (TFST)
Patient adherence / treatment discontinuation due to Adverse drug reactions (ADRs) / Serious adverse events (SAEs): | 24 weeks from randomization
  % of patients with treatment discontinuation due to specific ADRs (e.g. hand-foot syndrome, diarrhea, stomatitis, fatigue, hypertension)
Treatment Emergent Adverse Events according to CTC 4.03: | 24 weeks from randomization
  * Frequency/incidence, severity, percentage reduction, time-to-event of ADRs, AEs and specific TEAEs (e.g. hand-foot syndrome, diarrhea, stomatitis, fatigue, hypertension)
  * change of grade 3/4 ADRs
Assessment of comorbidities | at inclusion
  Charlson Comorbidity Index (CCI)

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Grünwald, Prof. Dr., Principal Investigator — Universitätsklinikum Essen
Locations (22):
- Germany (22):
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg, Bavaria
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Universitätsmedizin Göttingen, Göttingen, Lower Saxony
  - Universitätsklinikum Essen (AöR), Essen, Nordrhein-Westphalen
  - Hämatologisch-Onkologische Praxis Stolberg, Stolberg, North Rhine-Westphalia
  - Krankenhaus Barmherzige Brüder Trier, Trier, Rhineland-Palatinate
  - Universitätsklinikum Magdeburg A.ö.R., Magdeburg, Saxony-Anhalt
  - Urologische Arztpraxis Dr. Ralf Eckert, Wittenberg, Saxony-Anhalt
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Klinikum St. Marien Amberg, Amberg
  - Onkologisches Versorgungszentrum, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - BAG Onkologische Gemeinschaftspraxis, Dresden
  - Gemeinschaftspraxis Dr. med. Johannes Mohm Dr. med. Gabriele Prange Krex Fachärzte für Innere Medizin Hämatologie und Internistische Onkologie, Dresden
  - MVZ für Hämato/Onkologie Essen gGmbH, Essen
  - MVZ Onkologische Kooperation Harz, Goslar
  - Medizinische Hochschule Hannover, Hanover
  - Tagesklinik Landshut Hämatologie, Onkologie Palliativmedizin, Landshut
  - Klinikum Nürnberg 5. Medizinische Klinik, Nuremberg
  - Wissenschaftskontor Nord GmbH & Co KG, Rostock
  - Onkologische Schwerpunktpraxis, Singen
  - MVZ Kloster Paradiese GbR/Onkologiezentrum Soest, Soest

IPD SHARING:
Plan to Share IPD: No